CLINICAL TRIAL: NCT00200343
Title: A 24-week Multicenter Double-blind Control Trial With Ursodeoxycholic Acid in Patients With Chronic Hepatitis C
Brief Title: Efficacy and Safety Study of Ursodeoxycholic Acid to Treat Chronic Hepatitis C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MT711-01
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2011-11-07 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic hepatitis C, Ursodeoxycholic acid
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ursodeoxycholic Acid

ARMS (3):
- Ursodeoxycholic acid 150mg / day (Experimental)
  Interventions: Drug: Ursodeoxycholic acid 150mg / day
- Ursodeoxycholic acid 600mg / day (Experimental)
  Interventions: Drug: Ursodeoxycholic acid 600mg / day
- Ursodeoxycholic acid 900mg / day (Experimental)
  Interventions: Drug: Ursodeoxycholic acid 900mg / day

INTERVENTIONS:
Drug: Ursodeoxycholic acid 150mg / day — Ursodeoxycholic acid, 150mg/ day, three times a day at meals
  Arms: Ursodeoxycholic acid 150mg / day
Drug: Ursodeoxycholic acid 600mg / day — Ursodeoxycholic acid, 600mg/ day, three times a day at meals
  Arms: Ursodeoxycholic acid 600mg / day
Drug: Ursodeoxycholic acid 900mg / day — Ursodeoxycholic acid, 900mg/ day, three times a day at meals
  Arms: Ursodeoxycholic acid 900mg / day

SUMMARY:
This study is a 24-week multicenter, randomized, double-blind control trial with ursodeoxycholic acid (UDCA) in patients with chronic hepatitis C in Japan. The primary objectives of this study are to verify the superiority of efficacy of UDCA 600 or 900mg/day to that of 150mg/day and the safety of UDCA treatment.

DETAILED DESCRIPTION:
This study is a 24-week multicenter, randomized, double-blind control trial with ursodeoxycholic acid (UDCA) in patients with chronic hepatitis C in Japan. The primary objectives of this study are to verify the superiority of efficacy of UDCA 600 or 900mg/day to that of 150mg/day and the safety of UDCA treatment. The primary endpoint was percent changes of serum alanine aminotransferase(ALT) levels at 24-week of administration compared to pre-administration levels and secondary endpoints, serum aspartate aminotransferase(AST) and gamma-glutamyltranspeptidase(gamma-GTP) levels. Further, changes of bile acid composition and HCV-RNA levels at 24-week of administration were examined.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have a clinical diagnosis to apply the conservative medication for chronic hepatitis C.
2. Serum alanine aminotransferase levels measured at 4-week before the initiation of treatment must be over 61 IU/mL.
3. Subject's age must be 20 years or older.

Exclusion Criteria:

1. Subject who received a treatment of antiviral agents (interferon) within 20 weeks before the start of 8-week observation period
2. Subject who received a treatment of corticosteroids, immunosuppressive drugs, glycyrrhizic acid, cholestyramine or other drugs which could interfere with hepatic function during 8-week observation period.
3. Subject with decompensated cirrhosis
4. Subject infecting with other hepatic virus
5. Subject receiving a treatment for autoimmune disease, alcohol or drug-induced hepatic disorder, neoplasia, hepato-cholangiolar disease, fulminant hepatitis or peptic ulcer
6. Subject who require hospitalization for complications of the heart, kidney or pancreas
7. Pregnancy
8. Alcoholics
9. Alcohol intake more than 27 ml/day
10. Subject who involved in other clinical trial within 4 weeks before the start of observation period
11. Subject with a history of sensitivity to ursodeoxycholic acid or bile acid-products

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 596 (Actual)
Dates: Start 2002-07; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Overall Officials: Masao Omata, MD, Study Chair — Department of Gastroenterology, University of Tokyo
Locations (1):
- Department of Gastroenterology, University of Tokyo, Hongo, Bunkyo-ku, Tokyo, Japan

REFERENCES:
- [Result] Omata M, Yoshida H, Toyota J, Tomita E, Nishiguchi S, Hayashi N, Iino S, Makino I, Okita K, Toda G, Tanikawa K, Kumada H; Japanese C-Viral Hepatitis Network. A large-scale, multicentre, double-blind trial of ursodeoxycholic acid in patients with chronic hepatitis C. Gut. 2007 Dec;56(12):1747-53. doi: 10.1136/gut.2007.120956. Epub 2007 Jun 15. PMID 17573387

RESULTS

PARTICIPANT FLOW:
Groups:
- 150mg / Day: ursodeoxycholic acid, 150mg/day, three times a day at meals
- 600mg / Day: ursodeoxycholic acid, 600mg/day, three times a day at meals
- 900mg / Day: ursodeoxycholic acid, 900mg/day, three times a day at meals
Period: Overall Study
Arm/Group | 150mg / Day | 600mg / Day | 900mg / Day
Started | 199 | 200 | 197
Completed | 183 | 192 | 184
Not Completed | 16 | 8 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 150mg / Day | 600mg / Day | 900mg / Day | Total
Number analyzed (Participants) | 195 | 198 | 193 | 586
Age, Continuous [Mean (Standard Deviation); unit: years] — 10 patients were excluded from analysis population due to luck of sufficient data.
  years | 58.0 (12.2) | 57.7 (12.0) | 59.8 (10.1) | 58.4 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 81 | 70 | 249
  Male | 97 | 117 | 123 | 337

OUTCOME MEASURES:

1. Primary Outcome: Alanine Aminotransferase at Baseline
Time Frame: 0 week
Population: 10 patients were excluded from analysis population due to luck of sufficient data.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | 150mg / Day | 600mg / Day | 900mg / Day
Number analyzed (Participants) | 195 | 198 | 193
IU/L | 109.2 (49.7) | 106.3 (59.4) | 110.6 (57.3)

2. Secondary Outcome: Aspartate Aminotransferase at Baseline
Time Frame: 0 week
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | 150mg / Day | 600mg / Day | 900mg / Day
Number analyzed (Participants) | 195 | 198 | 193
IU/L | 84.0 (39.1) | 82.4 (41.8) | 85.2 (45.0)

3. Secondary Outcome: Percentage Change of Aspartate Aminotransferase From Baseline at Week 24
Description: Percentage change=[(measured value at Week 24 - measured value at baseline)/measured value at baseline]*100
Time Frame: 24 weeks (from baseline to Week 24)
Measure: Median (Full Range); unit: Percentage of change
Arm/Group | 150mg / Day | 600mg / Day | 900mg / Day
Number analyzed (Participants) | 195 | 197 | 192
Percentage of change | -13.6 [-74.2 to 347.2] | -25.0 [-82.7 to 72.5] | -29.8 [-79.0 to 1026.1]

4. Secondary Outcome: Gamma-glutamyl Transpeptidase at Baseline
Time Frame: 0 week
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | 150mg / Day | 600mg / Day | 900mg / Day
Number analyzed (Participants) | 195 | 198 | 193
IU/L | 87.5 (73.0) | 82.4 (62.2) | 85.9 (66.3)

5. Primary Outcome: Percentage Change of Alanine Aminotransferase From Baseline at Week 24
Description: Percentage change=[(measured value at Week 24 - measured value at baseline)/measured value at baseline]*100
Time Frame: 24 weeks (from baseline to Week 24)
Population: percentage change=[(measured value at Week 24 - measured value at baseline)/measured value at baseline]*100
Measure: Median (Full Range); unit: Percentage of change
Arm/Group | 150mg / Day | 600mg / Day | 900mg / Day
Number analyzed (Participants) | 195 | 198 | 193
Percentage of change | -15.3 [-80.7 to 375.9] | -29.2 [-88.3 to 95.2] | -36.2 [-81.4 to 1696.9]

6. Secondary Outcome: Percentage Change of Gamma-glutamyl Transpeptidase From Baseline at Week 24
Description: Percentage change=[(measured value at Week 24 - measured value at baseline)/measured value at baseline]*100
Time Frame: 24 weeks (from baseline to Week 24)
Population: percentage change=[(measured value at Week 24 - measured value at baseline)/measured value at baseline]*100
Measure: Median (Full Range); unit: Percentage of change
Arm/Group | 150mg / Day | 600mg / Day | 900mg / Day
Number analyzed (Participants) | 195 | 198 | 193
Percentage of change | -22.4 [-74.6 to 145.9] | -41.0 [-81.1 to 153.1] | -50.0 [-80.1 to 213.9]

ADVERSE EVENTS:
Time Frame: The reported adverse event data were collected for 24 weeks.
Arm/Group | 150mg / Day | 600mg / Day | 900mg / Day
Serious Adverse Events (participants affected / at risk) | 9/199 | 8/200 | 9/197
Other Adverse Events (participants affected / at risk) | 130/199 | 122/200 | 119/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 150mg / Day (N=199) | 600mg / Day (N=200) | 900mg / Day (N=197)
Colonic polyp (Gastrointestinal disorders) | 2 | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Appendicitis perforated (Gastrointestinal disorders) | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia NOS (Gastrointestinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0
Hepatic cirrhosis NOS (Hepatobiliary disorders) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hepatic neoplasm malignant NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 1
Renal neoplasm NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung cancer stage unspecified (excl metastatic tumours to lung) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Subarachnoid haemorrhage NOS (Nervous system disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Lumbar spinal stenosis (Nervous system disorders) | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 150mg / Day (N=199) | 600mg / Day (N=200) | 900mg / Day (N=197)
Abdominal distention (Gastrointestinal disorders) | 3 | 4 | 3
Abdominal pain NOS (Gastrointestinal disorders) | 4 | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 3 | 5 | 6
Constipation (Gastrointestinal disorders) | 4 | 4 | 6
Diarrhoea NOS (Gastrointestinal disorders) | 9 | 12 | 15
Dyspepsia (Gastrointestinal disorders) | 3 | 2 | 3
Loose stools (Gastrointestinal disorders) | 1 | 6 | 5
Nausea (Gastrointestinal disorders) | 3 | 2 | 3
Stomach discomfort (Gastrointestinal disorders) | 3 | 3 | 6
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 7
Chest discomfort (General disorders) | 5 | 1 | 0
Malaise (General disorders) | 2 | 5 | 2
Oedema peripheral (General disorders) | 1 | 2 | 3
Nasopharyngitis (Infections and infestations) | 51 | 49 | 52
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 6 | 5
Hepatic neoplasm malignant NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 6 | 1 | 3
Headache (Nervous system disorders) | 6 | 6 | 6
Insomnia (Psychiatric disorders) | 4 | 2 | 2
Cystitis NOS (Renal and urinary disorders) | 6 | 0 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 4
Eczema (Skin and subcutaneous tissue disorders) | 2 | 2 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 3 | 4
Rash NOS (Skin and subcutaneous tissue disorders) | 2 | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other